CLINICAL TRIAL: NCT06806423
Title: Clinical and Radiographic Evaluation of Topical Vitamin D Application on Immediate Dental Implants: a Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Topical Vitamin D on Immediate Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Bassem M. Ayyad, Bassem M. Ayyad, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vit D on Dental Implants
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Immediate Dental Implant; Implant Osseointegration; Vitamin D; Tooth Extraction
Keywords: Immediate dental implants; Calcitriol; 1,25-dihydroxycholecalciferol; Osseointegration; Implant stability; Bone density; IDRISI Kilimanjaro software

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): 12 implants were placed immediately after teeth extraction.
  Interventions: Procedure: Immediate Dental Implant Placement without Adjunctive Treatments
- Vitamin D Group (Experimental): 12 implants were placed immediately after teeth extraction, combined with topical vitamin D gel application.
  Interventions: Procedure: Immediate Dental Implant Placement with Topical Vitamin D Gel Application

INTERVENTIONS:
Procedure: Immediate Dental Implant Placement without Adjunctive Treatments — Atraumatic extractions using periotomes and anterior forceps. Osteotomy was prepared with a standardized drilling sequence under copious irrigation. ROOTT R-line implants were selected based on socket dimensions. No topical vitamin D3 was applied. Implants were placed into fresh extraction sockets.
  Arms: Control Group
Procedure: Immediate Dental Implant Placement with Topical Vitamin D Gel Application — The same procedure as the control group, with the addition of sterile topical vitamin D3 (calcitriol) gel applied to both the implant surface and osteotomy site immediately before implant placement.
  Arms: Vitamin D Group

SUMMARY:
This study evaluates the clinical and radiographic outcomes of topical vitamin D application on immediate dental implants in patients undergoing single-rooted tooth extraction in the anterior mandibular region.

DETAILED DESCRIPTION:
This randomized clinical trial investigates the clinical and radiographic outcomes of topical vitamin D application on immediate dental implants in patients undergoing single-rooted tooth extraction in the anterior mandibular region. Osseointegration, the direct structural and functional connection between bone and implant surface, is a critical factor in implant success. Recent studies suggest that vitamin D3 plays a significant role in bone metabolism, promoting osteoblast differentiation and enhancing mineralization. The aim of this study is to evaluate whether the adjunctive use of topical vitamin D3 gel can improve implant stability, peri-implant soft tissue health, and bone density around immediate dental implants.

Surgical Protocol:

* All surgical procedures were performed under strict infection control protocols at the Faculty of Dentistry, Suez Canal University.
* Patients rinsed with 0.1% chlorhexidine (Hexitol antiseptic mouthwash) for one minute before the procedure.
* The perioral area was disinfected using 10% povidone-iodine (Betadine).
* Local anesthesia was administered using 4% articaine hydrochloride with 1:100,000 epinephrine (Artinibsa) via the infiltration technique.
* Atraumatic tooth extractions were performed using periotomes and anterior forceps, preserving the surrounding alveolar bone.
* The dimensions of the extraction socket and residual bone were evaluated using a periodontal probe to ensure compatibility with the implant size.
* Osteotomy preparation followed a standardized protocol using sequential drills at 950-1100 rpm with 35 Ncm torque under copious irrigation to prevent overheating and bone necrosis.
* Study Group: Sterile vitamin D3 (calcitriol) gel was applied to both the implant surface and the osteotomy site immediately before implant placement.
* Control Group: No additional adjuncts were applied before implant placement.
* ROOTT R-line implants were selected based on socket dimensions.
* Implants were inserted into fresh extraction sockets, and proper alignment was meticulously confirmed to ensure ideal positioning.

Postoperative and Follow-up Evaluations:

* Clinical Assessments:

  * Pain levels were measured using the Visual Analog Scale (VAS) on postoperative days 1, 3, and 7.
  * Probing depth and bleeding index were recorded at 3 and 6 months to assess peri-implant soft tissue health.
  * Implant stability was evaluated using the Osstell ISQ device at baseline, 3 months, and 6 months.
* Radiographic Assessments:

  * Standardized digital periapical radiographs were taken at baseline, 3 months, and 6 months to monitor bone density changes around the implants.
  * Bone density analysis was performed using IDRISI Kilimanjaro software, which measured grayscale values to provide quantitative bone density assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders.
2. Middle-aged adults (from 21 years to 40 years).
3. Healthy American Society of Anesthesiologists patients (ASA I).
4. Patients with teeth or roots indicated for extraction at the lower anterior region.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Patients with parafunctional or bad oral habits such as bruxism or smoking (more than 10 cigarettes per day).
3. Patients with bad oral hygiene.
4. Patients with severe periodontal diseases (severe vertical or horizontal bone loss).
5. Pathological changes or infections related to teeth indicated for immediate implant placement.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Implant Stability (ISQ) | Baseline, 3, and 6 months postoperatively
  Implant stability was measured using the Osstell ISQ device, providing precise, non-invasive, and objective assessments for monitoring osseointegration. A SmartPeg was securely attached to the implant, and a probe connected to the device was positioned at a right angle toward the implant. The Implant Stability Quotient (ISQ) was measured on a scale from 1 to 100, with values above 70 indicating high stability, 60-69 indicating medium stability, and values below 60 suggesting low stability. Stability was assessed immediately after surgery and then reassessed at 3 and 6 months.
Bone Density | Baseline, 3 and 6 months postoperatively
  Radiographic evaluations were conducted using direct digital periapical radiographs, captured with the KaVo Scan eXam™ One system and Rinn XCP device. Radiographs were taken immediately postoperatively, and at 3 and 6 months. Bone density around the implants was analyzed using IDRISI Kilimanjaro software, which measured grayscale values to quantify density. Bone density was quantified on a 255-point grayscale, with 0 representing black regions and 255 representing white regions. Two zones were assessed: the osseointegration zone adjacent to the implant and the surrounding bone. This approach provided precise monitoring of bone density changes over time.

SECONDARY OUTCOMES:
Peri-implant Probing Depth (PD) | 3 and 6 months postoperatively
  Peri-implant probing depth was measured to assess the soft tissue healing surrounding the implants. A periodontal probe was gently inserted into the space between the implant healing abutments and the soft tissue at six sites: mesio-buccal, buccal, disto-buccal, mesio-palatal, palatal, and disto-palatal. Measurements were taken at 3 and 6 months postoperatively. The depth, recorded in millimeters, provided a numerical index of peri-implant tissue health, with shallow depths indicating healthy tissues and deeper pockets suggesting potential peri-implant disease. This straightforward method allowed for a comprehensive evaluation of implant sites over time.
Bleeding Index (BI) | 3 and 6 months postoperatively
  The Bleeding Index was used to assess the soft tissue healing surrounding the implants. A periodontal probe was gently inserted into the space between the implant healing abutments and the soft tissue at six sites: mesio-buccal, buccal, disto-buccal, mesio-palatal, palatal, and disto-palatal. Measurements were taken at 3 and 6 months postoperatively. The presence or absence of bleeding at these sites served as an indicator of tissue health, with bleeding suggesting inflammation or compromised healing, and no bleeding indicating healthy soft tissues. This method provided valuable insights into the status of soft tissue healing around the implants.
Visual Analogue Scale for Pain (VAS) | Days 1, 3, and 7 postoperatively
  The VAS is a commonly used questionnaire for measuring pain intensity. It consists of a 10-centimeter horizontal line with endpoints labeled to represent the extremes of pain, typically "no pain" on the left and "unimaginably unspeakable pain" or similar descriptors on the right. Patients are asked to mark a point on the line that reflects their current level of pain. The distance in centimeters from the "no pain" end to the patient's mark provides a numerical value representing the severity of their pain, offering a simple and quantifiable method for pain assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem M. Ayyad, Principal Investigator — Suez Canal University
Locations (1):
- Oral & Maxillofacial Surgery Department, Faculty of Dentistry, Suez Canal University, Ismailia, Ismailia Governorate, Egypt